CLINICAL TRIAL: NCT07219875
Title: Virtual Reality Training Study
Brief Title: Training Reward Responsiveness Through Virtual Reality
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michelle Craske, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-22-0269
Record Dates: First submitted 2025-09-22; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Positive Affect; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Virtual Reality-Reward Training (eVR-RT) (Experimental): 13 sessions of positive VR immersion and positive memory specificity training exercises designed to savor rewarding features of immersion followed by memory specificity training exercises to savor rewarding features of autobiographical memory
  Interventions: Behavioral: Enhanced Virtual Reality-Reward Training (eVR-RT)
- Virtual Reality-Memory Training (VR-MT) (Active Comparator): 13 sessions of neutral VR immersion and neutral memory specificity training exercises, designed to train memory of objective non-emotional stimuli followed by memory exercises to neutral non-personal stories
  Interventions: Behavioral: Virtual Reality-Memory Training (VR-MT)

INTERVENTIONS:
Behavioral: Enhanced Virtual Reality-Reward Training (eVR-RT) — Participants will complete verbal recounting (present-tense, field perspective, positive details) and guided imaginal recounting of positive details for rewarding VR experiences and positive autobiographical memories.
  Arms: Enhanced Virtual Reality-Reward Training (eVR-RT)
Behavioral: Virtual Reality-Memory Training (VR-MT) — Participants will complete verbal recounting (past-tense, observer perspective, objective details) and guided imaginal recounting of neutral details for neutral VR experiences and neutral non-personal stories
  Arms: Virtual Reality-Memory Training (VR-MT)

SUMMARY:
The purpose of this study is to compare the effects of enhanced Virtual Reality-Reward Training (eVR-RT) with an active control condition, Virtual Reality-Memory Training (VR-MT), on positive affect and other clinical symptoms.

Enhanced VR-Reward Training is a novel intervention aimed at enhancing savoring of positive experiences among individuals with depression and low positive affect through guided imaginal recounting following immersion in positive VR experiences. The current study tests an enhanced version of this training using improved virtual reality technology.

Target enrollment is 80 participants with low positive affect, depression, and impaired functioning, who are at least 18 years old, who will be randomly assigned to 7 weeks of either enhanced Virtual Reality-Reward Training (VR-RT) or Virtual Reality-Memory Training (VR-MT). Participants will complete in-person VR sessions, laboratory assessments, self-report questionnaires as part of the study. A subset of 8 participants randomly assigned to VR-RT will complete fMRI scans and EMA surveys.

The total length of participation is around 3 months.

DETAILED DESCRIPTION:
Anhedonia, or loss of interest and pleasure in usual activities, has been relatively resistant to pharmacological and psychological treatments in the context of anxiety and depression. Newer treatments that focus upon positivity or reward sensitivity have shown promising results.

The purpose of the current randomized controlled trial is to compare the effects of Enhanced Virtual Reality-Reward Training (eVR-RT) with an active control condition, Virtual Reality-Memory Training (VR-MT), on positive affect and other clinical symptoms. Enhanced Virtual Reality-Reward Training is designed to augment reward sensitivity in individuals with depression and low positive affect. Targets include reward anticipation and initial response to reward. Specificity of target engagement is assessed by comparison with Virtual Reality-Memory Training, designed to improve memory.

Targets and clinical outcomes are assessed at Week 0 Assessment (Week 0) and either weekly or at mid-treatment (Week 7), post-treatment (1 week after Session 14), and follow-up (Week 12). Statistical models evaluate whether change in outcomes and change in target measures are greater as a result of enhanced Virtual Reality-Reward Training compared to Virtual-Reality-Memory Training and whether changes in target measures correlate with changes in outcome measures.

Target enrollment is 80 participants with low positive affect, depression, and impaired functioning, who are at least 18 years old, who will be randomized to enhanced Virtual Reality-Reward Training or Virtual-Reality Memory Training, each comprising 13 individual virtual reality training sessions over the course of 7 weeks.

Participants will complete laboratory tests and self-report questionnaires as part of the study. Total length of participation is around 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Fluent in written and spoken English
3. Meet all of the following dimensional score cutoffs:

   1. Score on the DASS-21 depression subscale must be ≥ 8
   2. Score on the PANAS-P of 27 or lower
   3. Score on the WSAS of ≥ 11

Exclusion Criteria:

1. Lifetime history of bipolar disorder, psychosis, mental retardation, or organic brain damage
2. Substance use disorder in the past 6 months
3. Current use of psychotropic medications
4. Currently pregnant or planning to become pregnant
5. Self-reported frequent motion sickness
6. Self-reported seizures within the last year and/or a diagnosis of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The Mood and Anxiety Symptoms Questionnaire - Anhedonic Depression Subscale (MASQ-AD) | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  Change in reported anhedonia (score range: 14-70), with higher scores indicating greater anhedonic symptom severity
Positive Valence Systems Scale (PVSS-21) | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  Change in reward anticipation, motivation, and consumption for rewards such as rewards such as food, physical touch, positive feedback, social interactions, hobbies and goals (score range: 21-105). Higher scores (e.g. 105) indicate higher reward responsiveness.

SECONDARY OUTCOMES:
Depression, Anxiety, and Stress Scales (DASS-21) | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  Reported symptoms of depression (score range: 0-21), anxiety (score range: 0-21), and stress (score range: 0-21), higher scores indicate higher severity and frequency.
Positive and Negative Affective Schedule (PANAS) | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  Change in reported positive affect and negative affect (score range for each scale: 10-50, higher scores indicate higher levels of positive affect or negative affect) and will be measured weekly.
Positive and Negative Affective Schedule (PANAS-X) | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  The PANAS-X is a comprehensive measure comprised of 60 items assessing positive affect and negative affect. The PANAS-X will be administered at each assessment point
Responses to Positive Affect Questionnaire (RPA) | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  Change in rumination and dampening (Score range: 17-68). Higher scores indicate greater rumination and dampening.
Work and Social Adjustment Scale (WSAS) | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  The WSAS is used to assess the degree of impairment of a) work activities b) social life and leisure activities, and c) family life and home responsibilities. The scale discriminates depressed or anxious individuals in primary care who differ in impairment. Participants must score a 10 or above as their total, overall score to be included in the study.
igroup Presence Questionnaire (IPQ) | Change from Week 0 assessment to Post-Assessment (Week 8).
  The IPQ is a measure of 14 items assessing the sense of present in a virtual environment. The IPQ will be administered at each assessment point besides baseline.
Memory Retrieval Task | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  Change in accuracy in recalling neutral memories. Participants verbally recall a neutral distant memory (i.e., a memory that occurred longer than 2 weeks ago but closer than 3 months ago) and neutral recent (i.e., within past week) memory, then provide a word and sentence cue for each, to be used in future assessment sessions. At post-treatment and follow-up, the participants will be reminded of their word and sentence cue and recall both memories again verbally.
Heart Rate Variability | Change from VR Session 1 (Week 1) to VR Session 13 (Week 7).
  Change in heart rate variability (HRV). Data will be collected through actigraphy during session 1, 7, and 14. These data will be collected via a polar heartbeat monitor and actigraphy watch pairing. Actigraphy will be collected while the participant watches both VR scenes, the VR recall, and either the personal memory recall (eVR-RT) or the short story recall (VR-MT).
State Affect | Change from VR Session 1 (Week 1) to VR Session 13 (Week 7).
  A Visual Analogue Scale for Affect will be completed throughout the VR session, which assesses state affect before and after VR scenes and recountings. Higher scores (score range: 1-9) indicate higher affect.
Change in reward-relevant neural activity | Change from Week 0 Assessment to Post Assessment (Week 8)
  In a subset of 8 reward participants, the neural measure of reward-relevant neural reactivity including the ventral striatum and the medial orbitofrontal cortex (measured by fMRI) to assess change in reward processing from week 0 assessment to post-treatment. First-level voxel-wise z-statistics will be generated, contrasting reward anticipation (i.e., Win $0.50, Win $5.00) vs nonreward (i.e., Win $0.00), loss anticipation (i.e., Lose $0.50, Lose $5.00) vs non-loss (i.e., Lose $0.00), outcome of gain vs no-gain, and outcome of loss vs no-loss129.
Blood-Based Biomarkers | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  A small blood sample (approximately 1/8th teaspoon) will be collected at baseline, mid-treatment, post-treatment, and follow-up to measure peripheral inflammatory markers at these time points.
Depressive Symptoms Composite Score | Change from Week 0 assessment to Post-Assessment (Week 8). Change from Week 0 assessment to Follow-Up (Week 12).
  Change in a composite score of depressive symptoms including anhedonia (Measured by MASQ-AD), Depression (Measured by DASS-D), and low positive affect (Measured by PANAS).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States